CLINICAL TRIAL: NCT04342780
Title: Delayed Chemotherapy-induced Nausea: A Multi-center Prevalence Survey in Adult Oncology Patients in Clinical Practice
Brief Title: Prevalence of Delayed Chemotherapy Associated Nausea
Acronym: CINrate
Status: Completed | Type: Observational
Sponsor: Antje Koller (Other)
Collaborators: ZETUP St. Gallen (Unknown); Dr.-Hans-Altschüler-Stiftung (Unknown); University Medical Center Freiburg (Other); Spital Thurgau AG (Other)
Responsible Party: Sponsor-Investigator, Antje Koller, Principal Investigator, St.Gallen University of Applied Sciences
Organization: St.Gallen University of Applied Sciences (Other)
Other Study IDs: CINrate
Record Dates: First submitted 2020-03-25; First posted 2020-04-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: prevalence; chemotherapy-induced nausea and vomiting; oncology; suportive care
MeSH Terms: conditions — Vomiting; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the prevalence of delayed chemotherapy induced nausea in adult oncology patients in real clinical practice of day clinics.

DETAILED DESCRIPTION:
Chemotherapies are rated to have a high to minimal emetogenic potential in oncology patients. Their potential to induce delayed nausea is supposed to often be higher than their emetogenic potential. However, data on delayed chemotherapy-related nausea are scarce, which is problematic because nausea (a) has a large impact on patients quality of life and treatment decisions, (b) is often underestimated by health care professionals, (c) is less responsive to commonly used antiemetic medication, and (d) may even be different from rates that have been established in controlled clinical trials.

Therefore, the aim of this study is to assess the prevalence of delayed chemotherappy-induced nausea in adult oncology patients in dayclinics.

ELIGIBILITY:
Inclusion Criteria:

* first day of chemotherapy of a new cycle (any cycle)
* speak and write German
* sign the consent forms

Exclusion Criteria:

* cognitive or linguistic impairments that would significantly impede consent or participation (as assessed by the nurses in charge)
* accompanying radiotherapy;
* pre-existing nausea within three days before the start of the first chemotherapy in this cycle; and
* prior participation in CINrate (each person participates only once)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult oncology patients in dayclinics
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
delayed Nausea | Each patient: each days for 5 days after chemotherapy; recruitment: six weeks
  nausea that occurs 24 hours to 5 days after chemotherapy (100mm VAS in diary)

SECONDARY OUTCOMES:
acute nausea | Each patient: at day of chemotherapy at discharge from dayclinic; recruitment: six weeks
  nausea that occurs within 24 hours of chemotherapy (100mm VAS in diary)
acute and delayed vomiting | Each patient: each day for 5 days after chemotherapy; recruitment: six weeks
  vomiting that occurs within 5 days of chemotherapy (100mm VAS in diary)
adherence to antiemetics | Each patient: each day for 5 days after chemotherapy; recruitment: six weeks
  prescribed antiemetics compared with taken antiemetics; intake is calculated in % of the correct dose (dosing adherence) and in % of the dose at the right time (timing adherence)
antiemetic prescription | Each patient: at day of chemotherapy at discharge from dayclinic; recruitment: six weeks
  antiemetic medication that is prescribed
interference of nausea or vomiting with everyday life | Each patient: measured at day 5 after chemotherapy; recruitment: six weeks
  Functional Living Index Cancer (FLIE)
patient-related barriers to antiemetics | Each patient: measured at day 5 after chemotherapy; recruitment: six weeks
  Nausea and Vomiting Management Barriers Questionnaire (NVMBQ)

CONTACTS AND LOCATIONS:
Overall Officials: Antje Koller, Principal Investigator — Ostschweizer Fachhochschule St. Gallen
Locations (1):
- ZeTuP, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
we are planning to store anonymized data for further scientific use, however, this is depending on the vote of the ethical committee

REFERENCES:
- [Derived] Engst R, Glaus A, Moessner U, Ott S, Koller A. Delayed Chemotherapy-Induced Nausea - A Nurse-Led International Observational Study in Routine Oncology Practice (CINrate). SAGE Open Nurs. 2025 Dec 2;11:23779608251398116. doi: 10.1177/23779608251398116. eCollection 2025 Jan-Dec. PMID 41356791